CLINICAL TRIAL: NCT03215381
Title: An Open-Label Positron-Emission Tomography (PET) Study to Determine Brain Exposure of AZD1390 After Intravenous Administration of a Microdose [11C]AZD1390 to Healthy Volunteers
Brief Title: AZD1390 Administration of a Microdose [11C]AZD1390 to Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Karolinska Institutet, Quintiles IMS (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: D6940C00001
Record Dates: First submitted 2017-06-29; First posted 2017-07-12 (Actual); Last update posted 2018-02-26 (Actual); Status verified 2018-02

CONDITIONS: Healthy Volunteer Male Subjects
Keywords: Healthy Volunteer Male Subjects

STUDY DESIGN:
Masking Description: No Masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [11C]AZD1390 Microdose (Other): [11C]AZD1390 single dose not exceeding 10 ug by IV bolus
  Interventions: Drug: [11C]AZD1390

INTERVENTIONS:
Drug: [11C]AZD1390 — [11C]AZD1390
  Other Names: Radiolabeled AZD1390

SUMMARY:
This is an open-label, single centre exploratory study to analyse brain exposure of AZD1390 in healthy volunteer males.

DETAILED DESCRIPTION:
Up to 12 healthy male volunteers, 20 to 65 years of age will participate in the study. The study population chosen is sufficient to examine variability in pharmacokinetic and imaging measurements. All male volunteer subjects will have a baseline brain magnetic resonance imaging (MRI) for eligibility and anatomical delineation of brain regions to be applied in positron emission tomography (PET) image analysis. An arterial line will be inserted on day the healthy volunteer arrives for the administration of study drug and PET imaging (Day 1). The arterial line will be placed in the opposite arm than the one being used to administer the single intravenous microdose of [11C]AZD1390. Blood samples will be collected after the administration of microdose [11C]AZD1390 bolus injection and during the PET imaging procedure. The arterial line will be removed at the conclusion of the PET imaging study after the last blood sample has been collected. Standard institutional procedures will be followed for arterial line removal. The study will conclude with a telephone follow-up call within 7 business days after the PET measurement.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated, written informed consent prior to any study specific procedures.
* Healthy Male subjects, aged 20 to 65 years (inclusive).
* Subject should be healthy as determined by medical history, physical examination, laboratory parameters, ECG and brain MRI performed before administration of the investigational product.
* Subject should have a body mass index (BMI) between 18.0 and 30.0 kg/m2 and must weigh at least 50.0 kg and no more than 100.0 kg.
* Male subjects must be willing to adhere to true sexual abstinence or use condoms and spermicide (refer to Section 4.3); and refrain from donating sperm during the study and for 3 months plus 5 half-lives after the last administered radiolabelled infusion of [11C]AZD1390.
* Subject should be willing and able to participate in all scheduled evaluations, abide by study restrictions, and complete all required tests and procedures.

Exclusion criteria:

* Known or suspected neurological or behavioural disorders or symptoms that may interfere with the conduct or interpretation of the study, dementia (significant concomitant neurological disease are included under this category).
* Current significant major or unstable respiratory, heart, cerebrovascular, haematological, hepatic, renal, gastrointestinal diseases, or other major disease.
* Suffers from claustrophobia that limits the ability to undergo the scanning procedure.
* Subject has implanted metal devices or implants (MRI contraindications).
* Subject has received any concomitant medication or herbal medicine within 2 weeks prior to study drug administration.
* Subject has a negative Allen test in both hands at screening, unless brachial artery is used for arterial cannulation.
* Use of any anticoagulant within 30 days prior to study drug administration.
* Subject has previously participated in a PET imaging study.
* Central nervous system infarct, infection or focal lesions of clinical significance on brain MRI scan or abnormalities observed on the brain MRI that would interfere with image analysis
* As judged by the investigator, subject with unstable hypertension or symptomatic hypotension, history of pre-syncope or syncope due to orthostatic hypotension and/or induced by change of posture (orthostatic hypotension defined as 25 mmHg decrease in systolic and/or 15 mmHg).
* Presence of significant abnormalities on physical and neurological clinical examinations, vital signs, ECG and clinical chemistry, haematology, or urine analysis results at screening that may interfere with the study or present a safety risk to the study subject.
* History or positive results for a systemic infection (e.g. hepatitis B virus, hepatitis C virus, HIV, tuberculosis), including previous or on-going infectious or autoimmune disease at screening.
* History of alcohol or drug abuse or dependence (except nicotine) within 1 year prior to screening and/or urine drug screen positive for drug abuse.
* Prolonged QTcF >450 ms or family history of long QT syndrome.
* History of severe allergy/hypersensitivity or ongoing clinically significant allergy/hypersensitivity, as judged by the investigator or history of hypersensitivity to drugs with a similar chemical structure or class to [11C]AZD1390.
* Judgment by the investigator of any other reason that would prohibit the inclusion of the subject in the study.

Ages: 20 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2017-10-10 (Actual); Primary Completion 2018-02-19 (Actual); Study Completion 2018-02-19 (Actual)

PRIMARY OUTCOMES:
Brain distribution of AZD1390 | up to 2 hours post dose
  To assess if 11C AZD1390 crosses the blood brain barrier in healthy volunteers

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No